CLINICAL TRIAL: NCT02071472
Title: Evaluation of the Impact of an Electronic Pharmaceutical Record Used for Medication Reconciliation by a Pharmacist Associated to the Anesthesiologist Consultation
Brief Title: Electronic Pharmaceutical Record Used for Medication Reconciliation by a Pharmacist Associated to the Anesthesiologist Consultation
Acronym: DP-CONCIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DCIC 13 16
Record Dates: First submitted 2013-11-28; First posted 2014-02-26 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP medication reconciliation (Experimental): medication reconciliation by a pharmacist using an electronic pharmaceutical record associated to the anesthesiologist consultation for planned surgery patients.
  Interventions: Other: DP medication reconciliation
- control (No Intervention): conventional anesthesiologist consultation for planned surgery patients

INTERVENTIONS:
Other: DP medication reconciliation
  Arms: DP medication reconciliation

SUMMARY:
The objective is to evaluate the impact of an electronic pharmaceutical record used for medication reconciliation by a pharmacist associated to the anesthesiologist consultation

Experimental intervention:

medication reconciliation by a pharmacist using an electronic pharmaceutical record before the anesthesiologist consultation for planned surgery patients. The clinical pharmacist communicates the recommendations regarding the drug therapy to the anesthesiologist orally and using a specific formulary.

Control intervention:

Conventional anesthesiologist consultation for planned surgery patients.

DETAILED DESCRIPTION:
Anesthesiology consultation is mandatory in France for planned surgery. It is part of the concept of anesthesia safety. The main goal is to assess the anesthetic and surgical risk including clinical and drug features likely to interfere with the anesthesia. The medication reconciliation is a central part of this consultation especially in order to assess the allergic risk and hemostasis disorders.

However, access to comprehensive and reliable data concerning the consumption of health products by the patient represents a major challenge. The "Dossier Pharmaceutique" (DP) is an electronic pharmaceutical record including medications (prescribed medications, over the counter medications, complementary and alternative medicines) delivered by community pharmacists over a four month period. Hospital pharmacists have access to the DP of hospitalized patients in order to improve the quality of the medication reconciliation. These informations regarding medication of the patients will be shared with anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* patient coming for anesthetics consultation before a planned surgery
* age above18
* available electronic pharmaceutical record (DP)
* at least one medication prescribed before hospital admission

Exclusion Criteria:

* Minor patients ou majors protected by law
* Not speaking French patient
* Person who are not free by law or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1076 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-10 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a potential or documented adverse drug event collected by using trigger tool method | within the first 30 days after surgery

SECONDARY OUTCOMES:
Number of medications reported by the anesthesiologist in the medical record | winthin 2 to 4 weeks between anesthesiogist consultation and surgery

OTHER OUTCOMES:
Number of participants with a documented adverse drug event over the perioperative period | within the first 30 days after surgery
Demographic, clinical and therapeutic characteristics of all included participants | at inclusion
Number of participants having an electronic pharmaceutical record (DP) open | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierrick BEDOUCH, PharmD, PhD, Study Chair — University Hospital, Grenoble
Locations (1):
- Pharmacy Department - University Hospital of Grenoble, Grenoble, Isère, France

REFERENCES:
- [Derived] Chapuis C, Bosson JL, Bardet JD, Lepelley M, Sourd D, Roustit M, Allenet B, Chanoine S, Albaladejo P, Bedouch P. Electronic pharmaceutical record for best possible medication history at preoperative evaluation to prevent postoperative adverse events: a quasi-experimental study. BMJ Open Qual. 2025 Mar 3;14(1):e003022. doi: 10.1136/bmjoq-2024-003022. PMID 40032596